CLINICAL TRIAL: NCT04975230
Title: Sleep, Glycemia, and Self-Management in Young Adults With Type 1 Diabetes
Brief Title: Self-Management in Young Adults With Type 1 Diabetes
Acronym: SLEEPT1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20201829; K99NR018886 (NIH); R00NR018886 (NIH)
Record Dates: First submitted 2021-07-09; First posted 2021-07-23 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Young Adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Behavioral: Sleep self-management
Who Masked: Participant
Masking Description: Both conditions will receive time-balanced sessions with the study team. Participants will not be told whether in the experimental condition or the condition delivering usual care until after the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Self-Management (Experimental): The Sleep Self-Management Intervention involves an initial 50-minute face-to-face interactive session in a private location. Participants are asked to extend time in bed by 1 hour and consistently maintain the extension on both weekends and weekdays. Bedtimes and waketimes will be assessed to ascertain which time is most modifiable for the participant's lifestyle and routine. There will be weekly follow-ups and in-person 3-week booster sessions. Sleep reports generated by the actigraphy will be shared with participants with brief action planning and goal setting to address progress towards goal achievement. A need to revise plans for future weeks will be the booster sessions' major goal.
  Interventions: Behavioral: Sleep Self-Management
- Diabetes Self-Management Education (No Intervention): The Attention Control arm will receive Diabetes Self-Management Education at the initial consultation visit via in-person contact at T1. There will be weekly follow-ups and in-person 3-week sessions. A Diabetes Self-Management Tracking Form will be used to monitor the weekly acquisition of information and plans for the 6-week intervention and at the 3-month and 6-month data points.

INTERVENTIONS:
Behavioral: Sleep Self-Management — Intervention delivered by a sleep coach will include 1) initial in-person 50 min consultation; 2) brief 5 min weekly follow ups in a format TBD; and 3) in-person 30 min booster sessions every 3 weeks (total 13 sessions).
  Arms: Sleep Self-Management

SUMMARY:
Type 1 Diabetes (T1D) affects 1.6 million Americans, and only 14% of young adults age 18-25 years achieve glycemic targets (glycosylated hemoglobin A1C <7.0%). Achieving glycemic targets is associated with reduced risk for both micro-and macrovascular complications, better neurocognitive function, and better diabetes quality of life. In lab studies, sleep deprivation led to impaired glucose tolerance and insulin sensitivity in adults without chronic condition and in one study of adults with T1D. Extending sleep in natural environments contributes to improved insulin sensitivity and glucose levels, neurocognition, and psychological symptoms in young adults without chronic conditions. Modifiable dimensions of sleep health (appropriate sleep duration, stability, and timing) are associated with better glycemic control in adults with T1D. Therefore, improving sleep duration, stability, and timing may be potential therapeutic targets to improve glucoregulation and clinical outcomes (diabetes self-management, neurocognitive function, and symptoms) in this high-risk population.

The overall objective is to test and compare the effects of a cognitive-behavioral sleep self-management intervention (sleep extension and consistency in sleep timing) compared to an attention control condition (habitual sleep duration + diabetes self-management education) on improving sleep duration, stability, and timing, and glycemia (glycemic control and glucose variability) in short-sleeping young adults with T1D in a pilot randomized controlled trial.

DETAILED DESCRIPTION:
This is a two-arm randomized controlled trial, with participants assigned to either the Sleep Self-Management arm or the attention control arm (Diabetes Self-Management Education). The Sleep Self-Management condition involves an initial 50-minute face-to-face consultation with brief 5-10 minute weekly follow-ups in a format TBD by aim 1 (e.g., call, text, video conference) with 3-week booster sessions in person. The Sleep Self-Management intervention activities are provided in addition to "usual care."

ELIGIBILITY:
Inclusion Criteria:

* 1) Age range: from 18 to 26 years
* 2) Diagnosed with T1D for at least 6 months
* 3) No other major health problems (e.g., chronic medical condition or major psychiatric illness
* 4) Not currently participating in any intervention studies
* 5) Read/speak English
* 6) Have a most recent A1C or eA1C value ≥ 7%.

Exclusion Criteria:

* 1) Previous OSA diagnosis/high-risk sleep apnea
* 2) Current pregnancy
* 3) Night shift workers
* 4) Habitually sleep > 7 hours on work or school days.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Griggs, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals of Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was a single-center randomized controlled trial carried out at Case Western Reserve University between April 2022 and October 2023. Participants were recruited from Diabetes Specialty Clinics from University Hospitals Cleveland Medical Center.
Period: Overall Study
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Started | 21 | 18
Completed Intervention | 21 | 18
Completed (Completed Study) | 20 | 13
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Population: Thirty-Nine Participants Enrolled in Intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.95 (2.16) | 21.22 (2.39) | 21.08 (2.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 21 | 16 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 16 | 13 | 29
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Non-dominant Wrist-worn Actigraph to be Worn 24/7 (Spectrum Plus)
Description: Average sleep duration as assessed as the average minutes per night participants spent asleep over the 7-14 days preceding each time point (Change in sleep duration (longer sleep duration indicates improvement).
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Measure: Mean (Standard Error); unit: min per night
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
min per night | 18 (0.17) | -25.8 (0.17)
Statistical Analysis 1: Comparison: Sleep Self-Management vs Diabetes Self-Management Education; Test type: Other; p = 0.0227, Mixed Models Analysis; Cohen's D = 0.17, 95% CI 2-sided [-0.37 to 0.78], Standard Error of Mean 0.17

2. Primary Outcome: Time in Range 70-180 mg/dL
Description: Change in time in range 70-180mg/dL over the monitoring period (7-14 days). Continuous Glucose Monitor (CGM) data downloaded directly from each participant's existing or provided blinded Dexcom G6 [trademark]
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 19 | 14
percentage of time | 0.82 (4.35) | -0.35 (5.07)

3. Secondary Outcome: Diabetes Self-Management Questionnaire (27-item)
Description: Change in Diabetes Self-Management Questionnaire (DSMQ) scores. The DSMQ is a 27-item scale assessing behaviors and activities related to diabetes self-management. Each item is scored on a 4-point Likert scale from 0 (does not apply to me) to 3 (applies to me very much), and items scores are summed/transformed to a total score (range 0 to 10) reflecting overall diabetes self-management, with higher scores indicating better self-management skills (better outcome). This outcome represents the change in scores from baseline to post intervention. Diabetes self-management is an ongoing process where individuals actively manage their condition to maintain optimal blood sugar levels, prevent complications, and improve their overall quality of life.
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
score on a scale | 0 (1.40) | 0.44 (1.65)

4. Secondary Outcome: Paper-based Trail Making Test Parts A and B (Executive Function)
Description: Change in executive function (lower scores indicate improvement). The Trail Making Test (TMT) consists of two parts, A and B, which assess performance/cognitive function as the time taken to complete each part in seconds. In Part A, numbered circles (1-25) are connected in ascending order as quickly as possible. In Part B, circles are connected in ascending order with the added task of alternating between numbers and letters (1-A-2-B, etc.). Both parts are summed and scored based on the time taken to complete the task, with higher scores (longer time) indicating greater cognitive impairment.
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Population: intention to treat analysis - baseline values carried forward.
Measure: Mean (Standard Error); unit: time in seconds
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
time in seconds | -2.93 (0.79) | -0.92 (0.84)

5. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression Short Form
Description: Change in general distress (lower scores indicate improvement). The Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression Short Form is an 8-item instrument to assess depression symptoms. Each item is scored on a 5-point Likert scale from 1 (Never) to 5 (Always). Total raw scores range from 8-40 with higher scores indicating greater depressive symptoms.
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Population: Intention to treat, baseline values carried forward
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
score on a scale | 1.17 (2.06) | -0.34 (2.41)

6. Secondary Outcome: Diabetes Distress Scale (17-item)
Description: Change in diabetes distress (lower scores indicate improvement). The Diabetes Distress Scale (DDS) is a 17-item tool to measure emotional distress as experienced by individuals living with diabetes. Each item is scored on a 6-point Likert scale from 1 (Not a Problem) to 6 (A Very Serious Problem) with a total score range of 17-102
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Population: intention to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
score on a scale | -3.01 (3.03) | -2.22 (2.35)

7. Secondary Outcome: Diabetes Symptom Checklist Revised (34-item)
Description: Change in diabetes physical symptoms (lower scores indicate improvement). The Diabetes Symptom Checklist Revised (DSC-R) is a 34-item checklist to assess type 2 diabetes symptom burden using a 5-point Likert scale ranging from 0 (Not at all) to 5 (Extremely) with a total score range of 0-170 where higher scores indicate increased symptom burden
Time Frame: From (T0) baseline through 12-week intervention period (T2) captured immediately post intervention period.
Population: intention to treat analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 21 | 18
score on a scale | 0 (0.08) | -0.13 (0.09)

8. Other Pre Specified Outcome: 10-Minute Psychomotor Vigilance Test on a PVT-192 Device
Description: Change in Psychomotor Vigilance Test (PVT) score. The PVT as administered by the PVT-192 device (Ambulatory Monitoring) measures reaction time to assess alertness as an effect of sleep deprivation. Reactions are measure in time by seconds, where lower time scores in seconds indicating greater levels of alertness.
Time Frame: From (T0) baseline through (T3) 90 days post intervention
Population: The 10-Minute Psychomotor Vigilance Test on a PVT-192 device could not be administered/analysis completed for any enrolled participant due to hardware malfunction and lack of manufacturer technical assistance. The manufacturer was unable to provide timely support due to pandemic-related constraints. Data is not available now nor will it be available in the future.
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: This was a minimal risk behavioral trial.
Arm/Group | Sleep Self-Management | Diabetes Self-Management Education
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04975230/Prot_001.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04975230/SAP_002.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04975230/ICF_003.pdf